CLINICAL TRIAL: NCT04847687
Title: Health Sciences University Bursa Yüksek Ihtisas Training and Research Hospital
Brief Title: Investigation of Hospitalisation Times and Mortality According to Drug Dose in Patients Given Systemic Methylprednisolone With a Pre-diagnosis of Covid-19 Pneumonia; Retrospective Study
Status: Completed | Type: Observational
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Seyhan Dülger,MD, Health Sciences University Bursa Yüksek İhtisas Training and Research Hospital, Bursa Yuksek Ihtisas Training and Research Hospital
Other Study IDs: 2011-KAEK-25 2021/03-02
Record Dates: First submitted 2021-04-13; First posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: COVID-19; Methylprednisolone; Pneumonia
Keywords: COVID-19; Methylprednisolone; Pneumonia
MeSH Terms: conditions — COVID-19; Pneumonia | interventions — Methylprednisolone

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1: Patients who are started on 1 mg/kg/day methylprednisolone. Demographic data of the patients, length of hospital stay, follow-up in intensive care unit and prognosis will be recorded.
  Interventions: Drug: methylprednisolone
- Group 2: Patients who are started on 250 mg/day methylprednisolone. Demographic data of the patients, length of hospital stay, follow-up in intensive care unit and prognosis will be recorded.
  Interventions: Drug: methylprednisolone

INTERVENTIONS:
Drug: methylprednisolone — Patients who are hospitalized with a pre-diagnosis of severe COVID-19 pneumonia and who are started on methylprednisolone will be divided into two groups according to the drug dose. Groups will be compared in terms of length of hospital stay, intensive care needs and prognosis.
  Other Names: COVID-19

SUMMARY:
Aim:There is still not enough data to determine methylprednisolone treatment timing, dosage, duration of use and indication in Covid 19 pneumonia. The aim of this study is to examine the relationship between drug dose and hospitalisation time and mortality rates in patients with pre-diagnosis of severe covid pneumonia and systemic methylprednisolone.

Materials and Methods: The demographic data, symptom durations, thorax CT findings, methylprednisolone dose and duration of treatment, hospitalisation times, intensive care hospitalizations of the patients who were initiated and hospitalized in the emergency department will be retrospectively recorded. Finally, the fate of the patients (such as discharge, referral, death) will be recorded.Statistical analysis will be conducted using the Statistical Package for Social Sciences (SPSS) (IBM Corp. Released 2015. IBM SPSS Statistics for Windows, Version 21.0. Armonk, NY: IBM Corp.) program.

DETAILED DESCRIPTION:
Covid 19 infection can progress with widespread inflammation and cytokine storm. Induced excessive cytokine release is associated with tissue damage in the lung. Severe inflammatory / oxidative stress response and severe lung injury secondary to ARDS may develop. Therefore, suppressing the proinflammatory response has a very important place in treatment. Methylprednisolone is classically an immune response suppressor, powerful anti-inflammatory drug and is used in the treatment of covid 19 severe infection. However, there is still not enough data to determine the treatment timing, dosage, duration of use and indication.

The aim of this study is to examine the relationship between drug dose and hospitalisation time and mortality rates in patients with pre-diagnosis of severe covid pneumonia and systemic methylprednisolone.

Materials and Methods: The demographic data, symptom durations, thorax CT findings, methylprednisolone dose and duration of treatment, hospitalisation times, intensive care hospitalisations of the patients who were initiated and hospitalized in the emergency department will be retrospectively recorded. Finally, the fate of the patients (such as discharge, referral, death) will be recorded.

In the treatment of severe Covid 19 pneumonia, methylprednisolone treatment is used in addition to antiviral treatment. However, there are insufficient data on the time to start this treatment, drug dose and duration of use in daily routine. With the results of our study, we hope that we can contribute to the dose, duration and timing of methylprednisolone use in the treatment of Covid 19 pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years of age who presented to our hospital's emergency clinic
* Patients with pre-diagnosis of severe covid pneumonia
* Patients starting methylprednisolone therapy.

Exclusion Criteria:

* <18 years
* Patients with a pre-diagnosis of mild or moderate Covid 19 pneumonia
* Patients not hospitalized in our hospital
* Pregnant patients with Covid 19 pneumonia
* Patients whose 5-methylprednisolone treatment was started in the emergency and discontinued in less than 3 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years of age who presented to our hospital's emergency clinic with a pre-diagnosis of severe covid pneumonia and who were started on methylprednisolone treatment
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
prognosis | died during hospitalisation
  The patient was died.
hospitalization time | days between hospitalisation and externalization or death
  Time elapsed after the patient is hospitalized until person is discharged or died.

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Yüksek İhtisas EAH, Bursa, Eyalet/Yerleşke, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Demographic data of patients, duration of haspitalization, need for intensive care and prognosis will be shared with all researchers.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The data will be used for 3 months after April 1, 2021.